CLINICAL TRIAL: NCT02885610
Title: A Phase IIb , Placebo-Controlled ,Multi-Center, Randomized, Double-Blind, Dose-explorating Trial of RC18,a Recombinant Human B Lymphocyte Stimulating Factor Receptor-Antibody Fusion Protein in Subjects With Systemic Lupus Erythematosus (SLE).
Brief Title: Study of RC18 Administered Subcutaneously to Subjects With Systemic Lupus Erythematosus(SLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C005 SLECLLI
Record Dates: First submitted 2016-08-26; First posted 2016-08-31 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Standard of Care; RC-18

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo Comparator (Placebo Comparator): Placebo SC plus standard therapy; placebo once weekly ,and total of 48 doses
  Interventions: Biological: Placebo plus standard therapy
- RC18 80 mg plus standard therapy (Experimental): RC18 80 mg/kg SC plus standard therapy RC18 80 mg SC once weekly X 48 doses
  Interventions: Biological: RC18 80 mg plus standard therapy
- RC18 160 mg plus standard therapy (Experimental): RC18 160 mg/kg SC plus standard therapy RC18 160 mg SC once weekly X 48 doses
  Interventions: Biological: RC18 160 mg plus standard therapy
- RC18 240 mg plus standard therapy (Experimental): RC18 240 mg/kg SC plus standard therapy RC18 240 mg SC once weekly X 48 doses
  Interventions: Biological: RC18 240 mg plus standard therapy

INTERVENTIONS:
Biological: Placebo plus standard therapy — Standard therapy comprises any of the following (alone or in combination): corticosteroids, antimalarials, non-steroidal anti-inflammatory drugs (NSAIDs), and immunosuppressive and immunomodulator therapy(i.e.,azathioprine,mycophenolate ,cyclophosphamide,methotrexate,leflunomide, Tacrolimus ,ciclosporin )
  Other Names: Standard therapy
  Arms: Placebo Comparator
Biological: RC18 80 mg plus standard therapy — Standard therapy comprises any of the following (alone or in combination): corticosteroids, antimalarials, non-steroidal anti-inflammatory drugs (NSAIDs), and immunosuppressive and immunomodulator herapy(i.e.,azathioprine,mycophenolate ,cyclophosphamide,methotrexate,leflunomide, Tacrolimus ,ciclosporin )
  Other Names: Standard therapy
  Arms: RC18 80 mg plus standard therapy
Biological: RC18 160 mg plus standard therapy — Standard therapy comprises any of the following (alone or in combination): corticosteroids, antimalarials, non-steroidal anti-inflammatory drugs (NSAIDs), and immunosuppressive and immunomodulator herapy(i.e.,azathioprine,mycophenolate ,cyclophosphamide,methotrexate,leflunomide, Tacrolimus ,ciclosporin )
  Other Names: Standard therapy
  Arms: RC18 160 mg plus standard therapy
Biological: RC18 240 mg plus standard therapy — Standard therapy comprises any of the following (alone or in combination): corticosteroids, antimalarials, non-steroidal anti-inflammatory drugs (NSAIDs), and immunosuppressive and immunomodulator therapy(i.e.,azathioprine,mycophenolate ,cyclophosphamide,methotrexate,leflunomide, Tacrolimus ,ciclosporin )
  Other Names: Standard therapy
  Arms: RC18 240 mg plus standard therapy

SUMMARY:
The purpose of this study is to initially access the safety and effectivity of RC18 combined with standard treatment and Placebo combined with standard therapy in subjects with Moderate to severe SLE, Besides ,to provide dose basis for follow-up clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Active SLE disease，and at least according with 4 of the 11 items of the American College of Rheumatology (ACR) criteria 1997.
* Age & Gender: Male or female between 18 and 65 years of age inclusive，and the sex ratio is not limited
* Signed informed consent form，willing or able to participate in all required study evaluations and procedures.
* SELENA-SLEDAI(Safety of Estrogens in Lupus Erythematosus National Assessment SLE Disease Activity Index) score ≥ 8 during the screening period.and if there is hypocomlement or the Anti-dsDNA score, SELENA-SLEDAI disease activity score should be at least 6 at screening .
* Autoantibody-positive
* on a stable SLE treatment regimen for at least 30 days prior to Day 1, which consisted of any of the following (alone or in combination): cortical hormone,anti-malarials,non-steroidal anti inflammatory drugs (NSAIDs),or any immunosuppressive and immunomodulator therapy(i.e.,azathioprine,mycophenolate ,cyclophosphamide,methotrexate,leflunomide, Tacrolimus ,ciclosporin ).

Exclusion Criteria:

* Severe lupus nephritis within two months(designed as:Urine protein>6g/24h or serum creatinine ( SCr）>2.5mg/dL or 221umol/L ) or needing for hemodialysis or recepting high dose cortical hormone ≥14 days( metacortandracin>100mg/d or equivalent)
* Central nervous system disease caused by SLE or non SLE within two months (including epilepsy， mental disease，organic encephalopathy syndrome，cerebrovascular accident, encephalitis, central nervous system vasculitis）;
* there are serious heart, liver, kidney and other important organs and blood, endocrine system diseases and medical history;

Evaluation criteria for severity :

1. Alanine aminotransferase（ALT）or aspartate aminotransferase (AST) ≥2 upper limit of normal (ULN);
2. Creatinine Clearance (Ccr)<30ml/min;
3. White Blood Cell Count(WBCs)<2.5x 10(9)/L;
4. hemoglobin<85g/L;
5. Platelets<50x 10(9)/L.

   * Have a historically active hepatitis or active hepatitis or medical history,hepatitis B :Patients with positive HBsAg are excluded.;Hepatitis C: Patients with hepatitis C antibody positive are excluded;
   * Immune deficiency, uncontrolled severe infection and patients with active or recurrent peptic ulcer;
   * Pregnant , lactating women and men or women who have birth plans in the past 12 months ;
   * Have a history of allergic reaction to human biological medicines.
   * Receipt of live vaccine within 1 month;
   * Have participated in any clinical trial in the first 28 days of the initial screening or 5 times half-life period of the study compound (taking the time for the elderly).
   * Have received treatment with B cell targeted therapy such as Rituximab or Epratuzumab etc.
   * Receipt of anti-tumor necrosis factor、interleukin receptor antagonist；
   * Receipt of IV immunoglobulin（IVIG）,prednisone>100mg/d more than 14 days or plasma exchange;
   * There are active infections (such as herpes zoster, human immunodeficiency virus (HIV) virus infection, active tuberculosis, etc.) during the screening period;
   * Patients have depression or the significant suicide ideation;
   * Investigator considers candidates not appropriating for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2015-12; Primary Completion 2019-06-11 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
SLE Responder Index (SRI) Response Rate | Week 48
  At Week 48, the percent of subjects with ≥ 4 point reduction from baseline in SELENA SLEDAI score and increasing no more than 0.3 points in PGA and no new BILAG A organ domain score or 1 new BILAG B organ domain scores compared with baseline at the time of assessment.

SECONDARY OUTCOMES:
Percent of subjects with ≥ 4 point reduction from baseline in SELENA SLEDAI score | Week 48

OTHER OUTCOMES:
Mean Change From Baseline in PGA | Week 48
Percent of Subjects Whose Average Prednisone Dose Has Been Reduced by ≥ 25% From Baseline or ≤ 7.5 mg/Day During Weeks 44 Through 48 | Week 44 through 48
Mean Change From Baseline in Serological Examination Index(IgG、IgA、IgM) CD19+、Anti-dsDNA 、Complent C3、C4 | week 48

CONTACTS AND LOCATIONS:
Overall Officials: Fengchun Zhang, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wu D, Li J, Xu D, Merrill JT, van Vollenhoven RF, Liu Y, Hu J, Li Y, Li F, Huang C, Wang G, Li X, Zhao J, Zhao D, Huang C, Liu H, Wei W, Shi G, Lu F, Zuo X, Bi L, Li Z, Wang X, Zhang M, Tie N, Li J, Mo H, Fang J, Bao C, Zhang F. Telitacicept in patients with active systemic lupus erythematosus: results of a phase 2b, randomised, double-blind, placebo-controlled trial. Ann Rheum Dis. 2024 Mar 12;83(4):475-487. doi: 10.1136/ard-2023-224854. PMID 38129117